CLINICAL TRIAL: NCT03552094
Title: World Mosquito Program Noumea - Human Sample Component
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Pasteur (Industry)
Collaborators: Institut Pasteur of New Caledonia (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2017-036
Record Dates: First submitted 2018-05-28; First posted 2018-06-11 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Arbovirus Infections
Keywords: Arbovirus
MeSH Terms: conditions — Arbovirus Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemochromatosis or polycythemia patients: Blood samples from hemochromatosis or polycythemia patients requiring therapeutic bleeding that are not used in medical applications.
  Blood bag (volume of blood: from 450 to 500 mL).
  Interventions: Other: Blood donations of hemochromatosis or polycythemia patients
- Healthy donors: Blood samples from healthy donors. Blood bag (volume of blood: from 450 to 500 mL).
  Interventions: Other: Blood donations of healthy donors

INTERVENTIONS:
Other: Blood donations of hemochromatosis or polycythemia patients — Blood samples are from blood donations of hemochromatosis or polycythemia patients requiring therapeutic bleeding that are not used in medical applications.
  Groups: Hemochromatosis or polycythemia patients
Other: Blood donations of healthy donors — Blood samples are from blood donations of healthy donors.
  Groups: Healthy donors

SUMMARY:
The dengue, Zika and chikungunya arboviruses represent potentially severe infections to which the New Caledonian population is exposed. In the absence of specific treatment or vaccine, vector control remains the method of choice to limit their spread. However, the traditional methods of prevention and vector control measure today face their limits: mosquito resistance to insecticides, difficulty of access and destruction of breeding areas... The World Mosquito Program Noumea project is based on the artificial colonization of the mosquito vector Aedes aegypti by the endosymbiotic bacteria Wolbachia, which reduces its ability to transmit arboviruses. The breeding of mosquitoes carrying the bacterium Wolbachia in the laboratories of the Institut Pasteur of New Caledonia requires the use of human blood samples for mosquito gorging.

The objective of the research is to generate, maintain and amplify Aedes aegypti Caledonian lineages carrying the Wolbachia bacteria for the planned insect release program in Noumea.

DETAILED DESCRIPTION:
The dengue, Zika and chikungunya arboviruses represent potentially severe infections to which the New Caledonian population is exposed. In the absence of specific treatment or vaccine, disease vector control remains the method of choice to limit their spread. However, the traditional methods of prevention and disease vector control must today face their limits: mosquito resistance to insecticides, difficulty of access and destruction of breeding areas... The World Mosquito Program Noumea project is based on the artificial colonization of the mosquito vector Aedes aegypti by the endosymbiotic bacterium Wolbachia, which reduces its ability to transmit arboviruses. The breeding of mosquitoes carrying the bacterium Wolbachia in the laboratories of the Institut Pasteur of New Caledonia requires the use of human blood samples for mosquito gorging.

The objective of the research is to generate, maintain and amplify Aedes aegypti Caledonian lineages carrying the bacterium Wolbachia for the planned insect release program in Noumea.

The establishment of Wolbachia in Aedes aegypti populations in Noumea should lead to the reduction of active transmission of dengue, Zika and chikungunya in the municipality.

ELIGIBILITY:
Inclusion Criteria:

* All adult hemochromatosis or polycythemia patients or healthy donors have given their written consent to participate in the study and for the collection of a blood sample.

Exclusion Criteria:

* Participation refusal
* Minor person
* Positive result by Reverse transcription polymerase chain reaction RT-PCR for arboviruses
* Invalid qualification of the blood donation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hemochromatosis or polycythemia patients requiring therapeutic bleeding that are not used in medical applications, and healthy donors.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-06-25 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Generation of Aedes aegypti Caledonian lineages carrying the Wolbachia bacteria | 36 months
  Generation of Aedes aegypti Caledonian lineages carrying the Wolbachia bacteria for the planned insect release program in Noumea by measuring the Aedes aegypti female gorging rate
Maintenance and amplification of Aedes aegypti Caledonian lineages carrying the Wolbachia bacteria | 36 months
  Maintenance and amplification of Aedes aegypti Caledonian lineages carrying the Wolbachia bacteria for the planned insect release program in Noumea by measuring the number of eggs per Aedes Aegypti female gorged

SECONDARY OUTCOMES:
Vector competence assessment of the different Aedes aegypti Caledonian lineages | 36 months
  Assessment of the vector competence for the dengue, Zika and chikungunya viruses of the different Aedes aegypti Caledonian lineages with or without Wolbachia bacteria carriage by measuring the transmissibility reduction of Aedes aegypti carrying Wolbachia for arboviruses

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Touzain, Principal Investigator — Hospital Center of New Caledonia; Myrielle Dupont-Rouzeyrol, Principal Investigator — Institut Pasteur of New Caledonia
Locations (1):
- Centre Hospitalier de Nouvelle-Calédonie, Nouméa, Nouvelle-Calédonie, France